CLINICAL TRIAL: NCT02290756
Title: A Community Based Implementation of a Low Cost Evidence-based Toolkit and Parenting Program for Improving Brain Development in Newborns
Brief Title: A Community Based Implementation of a Toolkit and Parenting Program for Improving Brain Development in Newborns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Grand Challenges Canada (Other); Centre for Global Public Health Pakistan (Other)
Responsible Party: Principal Investigator, Dr. James F. Blanchard, Center Director, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H2014:301
Record Dates: First submitted 2014-10-21; First posted 2014-11-14 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Infant Development
Keywords: Early child development; Link Workers; Community Birth attendants; Parenting Program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parenting program and toolkit (Active Comparator): The intervention arm of the study will have the low cost evidence based toolkit delivered to the the pregnant women for the duration of their pregnancy and the parenting program delivered to the newborn for 12 months.
  Interventions: Behavioral: Parenting Program; Behavioral: Low cost evidence based toolkit
- Control- toolkit (Other): The control arm of the study will only have the low cost evidence based toolkit delivered to the the pregnant women for the duration of their pregnancy.
  Interventions: Behavioral: Low cost evidence based toolkit

INTERVENTIONS:
Behavioral: Parenting Program — The parenting program is an early childhood stimulation program aimed at newborns from their neonatal period till infancy. The implementation of the parenting program will be conducted through the link workers and parents of the newborns.
  Arms: Parenting program and toolkit
Behavioral: Low cost evidence based toolkit — The aim of providing the toolkit is to ensure that all pregnant women in the project are provided the requisite care needed from the antenatal period till delivery to limit complications and insults (both mother and especially the neonate) that can occur during pregnancy, delivery and post partum in both the mother and child. The contents of the toolkit will include:
  1. Clean delivery kit, aspiration bulb, bag and mask, Chlorhexidine, Misoprostol, Nutritional supplements (Iron and folic acid, awareness about breastfeeding) and IEC materials
  2. Trainings for Birth Attendants and Link workers on aspiration and hypothermia management techniques, use of bag and mask APGAR (also to parents), cord care, basic pregnancy and newborn care information

SUMMARY:
The investigators propose to develop and test the efficacy of a low cost evidence based toolkit aimed at improving brain development among newborns a rural setting of Pakistan. The toolkit will include a safe delivery kit, nutritional supplementation, and trainings on cord care, hypothermia management, aspiration and bag and mask techniques and APGAR score calculation. A simple, home-based parenting program will also be implemented that will teach parents tools that provide stimuli for brain and cognitive development in children. This parenting program covers Early Childhood Interventions for children at risk of developmental problems and covers developmental skill areas such as cognitive and fine motor, social and self-help and gross motor skills. Such an intervention package provides comprehensive care to families at the community level, with a minimal cost that can be scaled up. A new cadre of Link workers will be implemented who will provide mentoring and supportive supervision to Birth Attendants and will train parents in the stimulation program. The study will recruit 1080 pregnant women and their newborns.

DETAILED DESCRIPTION:
Intervention:

Through this project, two intervention packages will be implemented. Firstly the toolkit will be provided to all 1080 pregnant women recruited in both the intervention and control arm of the project. The aim of providing the toolkit is to ensure that all pregnant women in the project are provided the requisite care needed from the antenatal period till delivery to limit complications and insults (both mother and especially the neonate) that can occur during pregnancy, delivery and post partum in both the mother and child. The contents of the toolkit will include:

1. Gloves, Soap, a plastic sheet, a new razor blade, clean thread or narrow tape, cord clamp, aspiration bulb, bag and mask provision to the BAs, Chlorhexidine, Misoprostol, Nutritional supplements (Iron and folic acid, awareness about breastfeeding) and IEC materials
2. Trainings for Birth Attendants and Link workers on aspiration and hypothermia management techniques, use of bag and mask, APGAR (also to parents), cord care, basic pregnancy care and newborn care related information, danger signs during pregnancy, postpartum, for the newborn and during the neonatal and infancy.

The second intervention package will be the implementation of the parenting program through the link workers and parents to the newborns-followed monthly over a 12 month period and will be provided to 540 women only in the intervention arm of the study. The aim of this intervention is to improve brain development among newborns through the parenting program. The Curriculum for Child Development will be adapted to the community context and used. The curriculum will be developed in the first 6 months of the project and will be designed to include:

* Monthly lessons for the parents-this will include both group and individual sessions. The parents will have one group session and one follow-up individual session respectively.
* Training guides, materials/tools and diaries for the link workers to use to log the sessions The parenting program will be implemented by the Link Workers.

Project Implementation:

The project will proceed in two phases. In Phase 1 (first two months of the project) a community assessment will be conducted, operational plans finalized, development of tools, jobs aids, IEC materials, recruiting and trainings of the link workers and TBAs and other community based birth attendants. Furthermore, linkages with LHWs will be developed at this stage. The implementation toolkits will also be prepared, with all tangible elements procured in Pakistan.

Phase 2 will focus on implementing, monitoring and documenting interventions. In the first two months of Phase 2, pregnant mothers (who will be at the beginning of their second trimester) will be recruited in both arms of the study. Recruitment will be conducted by Birth Attendants and Link Workers through the listing of pregnant women developed in consultation with various formal and informal care providers in the community. Recruitment of women will be limited to these two months. Once recruited, the women will be followed for the duration of their pregnancy and through the first year of the newborn's life. Pregnant women will be provided services included in the toolkit including nutritional supplementation. In addition, the items of the toolkit that is essential for delivery such as the Clean Delivery Kit, Chlorhexidine and Misoprostol will be provided two months before the expected delivery date of each pregnant woman. Birth attendants trained through the project will deliver the home based deliveries that will take place in the communities. Referral networks will be established with referral health facilities in case of complications. Once the newborn is delivered, those in the intervention arm of the study will be provided the parenting program for the next 12 months. The newborns in the control arm will not be provided the parenting program, but will continue to receive the standard health care services provided through routine home-based visits of Lady Health Workers. Both the intervention and control groups will undergo assessments at varying times during the 12 month period when the parenting program will be implemented in the intervention group. These assessments will include assessing the parent-child interaction and conducting the home inventory test periodically starting from when the newborn is six months old. The Bayleys Scale for Infant Development-III will also be implemented on one year old infants (cognition, motor and language subtests) in both project arms.

ELIGIBILITY:
Inclusion Criteria:

1. Those pregnant women who are starting the second trimester of their pregnancy;
2. Those women who will continue to live in the community/village during the pregnancy period and until one year postpartum.

Exclusion Criteria:

1. Those pregnant women who appear to be, in the link worker's judgment, incapable of understanding the information provided about the study (e.g., mentally incapacitated, cognitively impaired etc.)
2. Not willing to participate in the study/unwilling to provide informed consent or the consent of their family.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1080 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Improvement in Bayleys Scale for Infant Development score | one time assessment at infant's 12 month birthday

SECONDARY OUTCOMES:
HOME inventory test | 2 assessments at 6 months birthday and 12 month birthday of the infant
  The Infant/Toddler (IT) HOME Inventory is designed for use during infancy (birth to age three). It is composed of 45 items clustered into six subscales: 1) Parental Responsivity, 2) Acceptance of Child, 3) Organization of the Environment, 4) Learning Materials, 5) Parental Involvement, and 6) Variety in Experience. Each inventory contains a group of scales to assess different aspects of the child's environment. Each scale contains a number of items that are scored according to a glossary. The HOME therefore provides a framework for interviewers to assess all aspects of the home environment, including parenting, that directly impact on the child.
Parent-Child Interaction assessment | 2 assessments at 6 months birthday and 12 month birthday of the infant
  This tool will consist of a checklist that will observe the different behaviors of the mother, while the child is given an object to play with. It looks at the mother's sensitivity to the child's needs. In addition, this questionnaire also observes the mother's effort to help a child to maintain interest level in that particular game.
  Another checklist aimed at observing the infant will be used to observe the infant's response to the game the mother wants to play with e.g, excitement and enjoyment like clapping etc. Observation of the child's communication towards the mother and the game will also be assessed, to see whether the response is positive, negative, and to see what effort the child makes to communicate.

CONTACTS AND LOCATIONS:
Overall Officials: James F Blanchard, MSc, Principal Investigator — University of Manitoba; Tahira E Reza, MSc, Principal Investigator — Centre for Global Public Health Pakistan
Locations (1):
- Center for Global Public Health, Islamabad, Pakistan